CLINICAL TRIAL: NCT02840682
Title: Outcomes of Neonatal Resuscitation in a Resource Limited Setting on the Thailand-Myanmar Border
Brief Title: Outcomes of Neonatal Resuscitation
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: SMRU1603
Record Dates: First submitted 2016-06-07; First posted 2016-07-21 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Neonatal Resuscitation
Keywords: resource limited setting; Thailand-Myanmar border

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this study is to describe mortality of newborns who received basic, advanced or no neonatal resuscitation immediately after birth at Shoklo Malaria Research Unit.

DETAILED DESCRIPTION:
This is a retrospective, descriptive study of hospital records will be conducted. The existing dataset of newborns of ≥28 weeks gestation delivered at Shoklo Malaria Research Unit clinics from January 2008 to December 2015 will be analysed.

In the dataset, 15224 newborns fulfill the inclusion criteria and therefore they will all be analysed with IBM SPSS Statistics 22 for Windows.

Descriptive statistics will be used to define: a) the proportion of newborns alive at 24 hours, 7 days, 28 days, and at 1 year, following resuscitation at SMRU birthing rooms and b) the number of newborns requiring basic and advanced resuscitation.

Measurements of correlation coefficient will be used to compare Shoklo Developmental test scores and developmental milestones attained at 1 year in resuscitated and non-resuscitated infants. The Pearson correlation coefficient will be used if the relationship between two variables is found to be linear.

Antenatal, perinatal and postnatal characteristics associated with neonatal resuscitation will be defined by logistic regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* Liveborn singletons birthed at SMRU
* ≥28 weeks gestation

Exclusion Criteria:

* Stillborn infants
* Liveborn infants birthed at home or in the Thai hospital
* Major congenital abnormalities

Max Age: 28 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All liveborn, singletons, ≥28 weeks gestation, birthed at SMRU, from 1 January 2008 to 31 December 2015 will be included.
Sampling Method: Non-Probability Sample
Enrollment: 15073 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-08-15 (Actual); Study Completion 2016-08-15 (Actual)

PRIMARY OUTCOMES:
Mortality 24 hours after birth of babies who received basic resuscitation | 24 hours
Mortality 24 hours after birth of babies who received advanced resuscitation | 24 hours
Mortality 24 hours after birth of babies who did not receive neonatal resuscitation | 24 hours

SECONDARY OUTCOMES:
Mortality at 7 days | 7 days
Mortality at 28 days | 28 days
Mortality at one year | 1 year
Proportion of live births requiring basic or advanced neonatal resuscitation. | 24 hours
Number of newborns who received basic resuscitation, as a proportion of all live births. | 24 hours
Number of newborns who received advance resuscitation, as a proportion of all live births. | 24 hours
Shoklo Developmental test scores at 1 year in infants who received basic or advanced neonatal resuscitation or no resuscitation. | up to 1 year of age
Month of achieved milestones (crawl, walk, talk) in in infants who received basic or advanced neonatal resuscitation or no resuscitation. | up to 1 year of age
characteristics of antenatal infant receiving neonatal resuscitation compared to non-resuscitated infants as assessed by physiological parameter | 24 hours
characteristics of perinatal infants receiving neonatal resuscitation compared to non-resuscitated infants as assessed by physiological parameter | 24 hours
characteristics of neonatal infants receiving neonatal resuscitation compared to non-resuscitated infants as assessed by physiological parameter | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Shoklo Malaria Research Unit, Mae Sot, Changwat Tak, Thailand

IPD SHARING:
Plan to Share IPD: Yes